CLINICAL TRIAL: NCT03646721
Title: A Phase 1b, Double-Blind, Placebo-Controlled, Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, PK and PD of DA-1241 in Healthy Male Subjects and Subjects With T2DM
Brief Title: A Study to Evaluate the Safety, Tolerability, PK and PD of DA-1241 in Healthy Male Subjects and Subjects With T2DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA1241_DM_Ib
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — DA-1241; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- [Part1] DA-1241 : 6 subjects in each cohort(Cohort 1-3) (Experimental): Subjects will participate in 1 of 3 cohorts consisting of 8 subjects per cohort. Within cohorts, subjects will be randomized to a ratio of 6:2 (DA-1241 to matching placebo).
  Interventions: Drug: DA-1241
- [Part1] Placebo : 2 subjects in each cohort(Cohort 1-3) (Placebo Comparator): Subjects will participate in 1 of 3 cohorts consisting of 8 subjects per cohort. Within cohorts, subjects will be randomized to a ratio of 6:2 (DA-1241 to matching placebo).
  Interventions: Drug: Placebo
- [Part2] DA-1241 : 15 subjects in each cohort(Cohort 4-6) (Experimental): Subjects will participate in 1 of 3 cohorts consisting of 25 subjects per cohort. Within cohorts, subjects will be randomized to a ratio of 3:1:1 (DA-1241 to matching placebo and active comparator).
  Interventions: Drug: DA-1241
- [Part2] Placebo : 5 subjects in each cohort(Cohort 4-6) (Placebo Comparator): Subjects will participate in 1 of 3 cohorts consisting of 25 subjects per cohort. Within cohorts, subjects will be randomized to a ratio of 3:1:1 (DA-1241 to matching placebo and active comparator).
  Interventions: Drug: Placebo
- [Part2] Sitagliptin : 5 subjects in each cohort(Cohort 4-6) (Active Comparator): Subjects will participate in 1 of 3 cohorts consisting of 25 subjects per cohort. Within cohorts, subjects will be randomized to a ratio of 3:1:1 (DA-1241 to matching placebo and active comparator).
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: DA-1241 — [Part1] Administration once daily for 28 days; Dose strength for each cohort (Cohort 1, 2 and 3) is planned as 50mg, 100mg and 200mg, respectively.
  [Part2] Administration once daily for 56 days; Dose strength for each cohort (Cohort 4, 5 and 6) is planned as 25mg, 50mg and 100mg, respectively.
  (Dose escalation and dose level decisions for subsequent cohorts will be made via interim dose escalation review meetings.)
  Arms: [Part1] DA-1241 : 6 subjects in each cohort(Cohort 1-3); [Part2] DA-1241 : 15 subjects in each cohort(Cohort 4-6)
Drug: Placebo — [Part1] Administration once daily for 28 days. [Part2] Administration once daily for 56 days.
  Arms: [Part1] Placebo : 2 subjects in each cohort(Cohort 1-3); [Part2] Placebo : 5 subjects in each cohort(Cohort 4-6)
Drug: Sitagliptin — [Part2] Administration of Sitagliptin 100mg once daily for 56 days.
  Arms: [Part2] Sitagliptin : 5 subjects in each cohort(Cohort 4-6)

SUMMARY:
This is a double-blind, placebo-controlled, multiple ascending dose study to evaluate the safety, tolerability, PK and PD of DA-1241 in healthy male subjects and subjects with T2DM

ELIGIBILITY:
<Part 1>

Inclusion Criteria:

1. Healthy male subjects
2. Age ≥ 18 to ≤ 70 years of age.
3. Body mass index (BMI) ≥ 18.5 to ≤ 29.9 kg/m2.
4. Non-diabetic, fasting plasma glucose (FPG) of < 100 mg/dL (measured with YSI at site; one repeat test is allowed)
5. HbA1c < 5.7 %
6. Non-smoker smoker, defined as: Non-smoker for >12 months (ie, subject has not smoked or used any tobacco product for the 12 months prior to the start of the study) confirmed by a negative nicotine/cotinine test.
7. Male subjects must be surgically sterile, or engaged with partners of non-childbearing potential, or if engaged with partners of childbearing potential, the subject and his partner must be willing to use contraceptive methods until 3 months after the last day of IP administration. Males must not donate sperms during the study and until 3 months after the last day of IP administration.
8. Upon review, agree to participate and sign informed consent

Exclusion Criteria:

1. Resting blood pressure (BP) > 140/90 mmHg or < 90/60 mmHg. Subjects BP may be re-checked.
2. Participation in an investigational drug/device study within 30 days or 5 half-lives within the last dose of any study drug, whichever is longer.
3. History of any serious adverse reaction or hypersensitivity to any of the investigational product components or medicinal products with similar chemical structure.
4. Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders or abnormalities, or other major systemic disease that, according to the investigator, would unduly risk the subject's safety or may impact the conduct of the study.
5. History of or acute significant gastrointestinal disorder (eg, peptic ulcers, severe GERD), gastric surgery, including surgical treatment for obesity (eg, bariatric surgery, gastric banding), gastric bypass or antrectomy or small bowel resection >20cm or any disorder that would interfere with the swallowing, absorption, distribution, metabolism and excretion of the investigational product. Surgery for appendicitis is acceptable.
6. Subject shows evidence of significant active neuropsychiatric disease, including taking prescription medication for such diseases (including anti-depressant /anti-anxiety medication),
7. Presence of clinically significant physical, laboratory, or ECG findings at Screening that, in the opinion of the Investigator, may interfere with any aspect of study conduct or interpretation of results, or may present a safety issue to that particular subject. (Laboratory results may be re-checked once on a separate day per Investigator discretion)
8. Long QT syndrome or family history of long QT syndrome or corrected QT interval (QTcF) > 450 ms at screening.
9. Liver function test results of AST and/or ALT ≥ 1.5 upper limit of normal (ULN).
10. Subject had a history of vaso-vagal syncope within 5 years.
11. History of any major surgery within 6 months.
12. History of any active infection, other than mild viral illness within 30 days prior to dosing.
13. Known history or positive test of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus type 1 (HIV-1) or 2 (HIV-2) antibody.
14. Subjects with a positive urine nicotine/cotinine dipstick test.
15. History of alcohol abuse as judged by the Investigator within approximately 1 year. Average weekly alcohol intake > 21 units/week or are unwilling to stop alcohol consumption from 24 hours prior to each dosing until discharged from the clinical research unit (CRU). Positive alcohol test at Screening. (One unit of alcohol equals about 250 mL of beer or lager, 100 mL of wine, or 35 mL of spirits).
16. History of illicit drug abuse, within approximately 1 year or evidence of current use as judged by the Investigator. Positive drug test, including marijuana, at Screening.
17. Donation or loss of > 500 mL of blood within 56 days.
18. Chronic use of over-the-counter or prescription medication within 7 or 14 days prior to dosing per Investigator's discretion (apart from vitamin/mineral supplements, occasional paracetamol, or birth control methods).
19. Unable to comply with the safety monitoring requirements of this clinical study or is considered by the investigator to be an unsuitable candidate for the study.

<Part 2>

Inclusion Criteria:

1. Male and female subjects with T2DM > 6 months.
2. Age ≥ 18 to ≤ 70 years of age.
3. Body mass index (BMI) ≤ 35 kg/m2.
4. On stable therapy with metformin monotherapy or metformin in combination with other oral antidiabetic drugs (OADs) ≥ 1 month. (OADs except metformin will be washed-out prior to the first dosing)
5. HbA1c ≥ 6.5 to ≤ 10%
6. Female and male subjects must agree to use highly effective methods of birth control until 120 days after the last day of IP administration, or must be surgically sterile or postmenopausal. Males must not donate sperm during the study and until 120 days after the last day of IP administration.
7. Upon review, agree to participate and sign informed consent.

Exclusion Criteria :

1. A subject who has acute proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy, especially autonomic neuropathy, as judged by the Investigator.
2. Recurrent major hypoglycemia or hypoglycemic unawareness or recent ketoacidosis, as judged by the Investigator.
3. Persistent blood pressure (BP) systolic or diastolic > 160/90 mmHg or < 90/60 mmHg. Subjects BP may be re-checked per site SOP. Treatment with stable doses of antihypertensive medication for 2 months prior to screening are allowed.
4. Pregnant or lactating women.
5. Participation in an investigational drug/device study within 30 days or 5 half-lives within the last dose of any study drug, whichever is longer.
6. History of any serious adverse reaction or hypersensitivity to any of the investigational product components or medicinal products with similar chemical structure.
7. Current use of any prescribed or non-prescribed drugs (other than current treatment for diabetes mellitus or birth control methods) that are known to interfere with glucose or insulin metabolism, including but not limited to oral corticosteroids, GLP-1 receptor agonists, monoamine oxidase (MAO) inhibitors, growth hormone, non-selective β-blockers and lipid lowering medication. Lipid lowering medications will be washed-out prior to the first dosing if subjects take medication for primary prevention.
8. History of administration or current use of thiazolidinediones (TZDs).
9. Chronic use of acetaminophen, as acetaminophen is not allowed during the CGMS periods in the study.
10. Unable to tolerate tape adhesive in the area of sensor placement.
11. Subject has any unresolved adverse skin condition in the area of sensor placement (eg, psoriasis, rash, Staphylococcus infection).
12. History of or acute significant gastrointestinal disorder (eg, peptic ulcers, severe GERD), gastric surgery, gastric bypass or antrectomy or small bowel resection or any disorder that would interfere with the swallowing, absorption, distribution, metabolism and excretion of the investigational product. Surgery for appendicitis is acceptable.
13. History of renal disease or abnormal kidney function tests at Screening (eGFR < 60 mL/min/1.73m2 as estimated using the MDRD equation).
14. Clinically significant abnormal laboratory test, in particular, elevated liver enzymes (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 2 times the upper limit of normal (ULN)). (Laboratory results may be re-checked once on a separate day per Investigator discretion)
15. Any history of heart disease, defined as symptomatic heart failure (New York Heart Association class III or IV), myocardial infarction, coronary artery bypass graft surgery, or angioplasty, unstable angina requiring medication, transient ischemic attack, cerebral infarct, or cerebral hemorrhage.
16. History of any clinically or active significant gastrointestinal, cardiovascular, hematological, psychiatric, renal, hepatic, pancreatic or neurological abnormality that could interfere with the safety or results of this study as judged by the Investigator.
17. Subject shows evidence of significant active neuropsychiatric disease. Subjects that are stable and controlled by stable doses of selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), antipsychotics and lithium for ≥ 6 months prior to screening are allowed.
18. Presence of clinically significant physical or ECG findings (eg, QTcF > 450 msec for males, QTcF > 470 msec for females, left bundle branch block (LBBB)) at Screening that, in the opinion of the Investigator, may interfere with any aspect of study conduct or interpretation of results, or may present a safety issue to that particular subject.
19. History of any major surgery within 6 months.
20. History of any active infection, other than mild viral illness within 30 days prior to the first dosing.
21. Known history or positive test of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus type 1 (HIV-1) or 2 (HIV-2) antibody.
22. Smoking > 10 cigarettes per day or equivalent use of any tobacco product (eg, nicotine patch) within 6 months prior to Screening. Subjects must be able to refrain from smoking during each in-house period.
23. History of alcohol abuse as judged by the Investigator within approximately 1 year. Average weekly alcohol intake > 21 units/week (males) and > 14 units/week (females) or are unwilling to stop alcohol consumption from 24 hours prior to each check-in for in-house and outpatient visits and throughout the in-house periods until discharged from the clinical research unit (CRU) and are unwilling to limit alcohol consumption during outpatient periods. Positive alcohol test at Screening. (One unit of alcohol equals about 250 mL of beer or lager, 100 mL of wine, or 35 mL of spirits).
24. History of illicit drug abuse, within approximately 1 year or evidence of current use as judged by the Investigator. Positive drug test, including marijuana, at Screening.
25. Donation or loss of > 500 mL of blood within 56 days.
26. Unable to comply with the safety monitoring requirements of this clinical study or is considered by the investigator to be an unsuitable candidate for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
12-lead ECGs | Throughout study duration, i.e., about 10 weeks (Part1) and about 14-16 weeks (Part2), respectively
  Change from baseline in QTcF (msec)
Blood pressure | Throughout study duration, i.e., about 10 weeks (Part1) and about 14-16 weeks (Part2), respectively
  Change from baseline in blood pressure (mmHg)
Heart rate | Throughout study duration, i.e., about 10 weeks (Part1) and about 14-16 weeks (Part2), respectively
  Change from baseline in heart rate (bpm)
Body temperature | Throughout study duration, i.e., about 10 weeks (Part1) and about 14-16 weeks (Part2), respectively
  Change from baseline in oral body temperature (°C)
Respiratory rate | Throughout study duration, i.e., about 10 weeks (Part1) and about 14-16 weeks (Part2), respectively
  Change from baseline in respiratory rate (bpm)
Physical examination | Throughout study duration, i.e., about 10 weeks (Part1) and about 14-16 weeks (Part2), respectively
  Incidence and severity of clinical findings on physical examination
Clinical laboratory testing | Throughout study duration, i.e., about 10 weeks (Part1) and about 14-16 weeks (Part2), respectively
  Incidence and severity of clinical laboratory abnormality
Adverse event | Throughout study duration, i.e., about 10 weeks (Part1) and about 14-16 weeks (Part2), respectively
  Incidence and severity of adverse event

SECONDARY OUTCOMES:
Maximum concentration of DA-1241 (Cmax) | Through the treatment period; 24 hours
Time of maximum plasma DA-1241 concentration (Tmax) | Through the treatment period; 24 hours
Area under the concentration-time curve (AUC) | Through the treatment period; 9 days
Apparent terminal elimination half-life (t½) | Through the treatment period; 9 days
Apparent total systemic clearance after oral administration (CL/F) | Through the treatment period; 9 days
Apparent volume of distribution (Vz/F) | Through the treatment period; 9 days
Accumulation ratio (Last dosing day AUCtau / First dosing day AUCtau) | Through the treatment period; 9 days
Amount of DA-1241 excreted unchanged in the urine in each collection interval(Ae) | Through the treatment period; 7 days
Cumulative amount of DA-1241 excreted unchanged in the urine (Cum Ae) | Through the treatment period; 7 days
Percentage fraction of DA-1241 excreted unchanged in the urine in each collection interval(Fe) | Through the treatment period; 7 days
Cumulative percentage fraction of DA-1241 excreted unchanged in the urine (Cum Fe) | Through the treatment period; 7 days
Renal clearance (CLR) | Through the treatment period; 7 days
Fasting Plasma Glucose (FPG) | Through the treatment period; 62 days
2h-Postprandial glucose | Through the treatment period; 56 days
Area under the measurements versus (vs) time curve(AUE) | Through the treatment period; 56 days
Incremental AUEs after meal (iAUE) | Through the treatment period; 56 days
Weighted mean glucose (WMG) | Through the treatment period; 56 days
Incremental WMG (iWMG) | Through the treatment period; 56 days
Fasting Insulin | Through the treatment period; 56 days
Glycated albumin | Through the treatment period; 56 days
HbA1c | Through the treatment period; 56 days

OTHER OUTCOMES:
Assessment of key metabolite(s) of DA-1241 | Through the treatment period; 41 days
  Key metabolite(s) of DA-1241 will be assessed in blood and urine.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Site, Chula Vista, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - High Point Clinical Trials Center, High Point, North Carolina
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No